CLINICAL TRIAL: NCT03978949
Title: Prevention of Radiotherapy Induced Enteropathy by Probiotics (PREP Trial): a Prospective, Randomized Controlled, Double Blinded, Single Center, Superiority Study
Brief Title: Prevention of Radiotherapy Induced Enteropathy by Probiotics (PREP)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Seok Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S2019-0657-0003
Record Dates: First submitted 2019-05-31; First posted 2019-06-07 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Radiotherapy; Toxicity; Diarrhea; Probiotics
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Two weeks prior to the start of radiation therapy, the probiotics is administered three times daily until the end of radiation therapy.
  Interventions: Drug: Bacillus Licheniformis
- Placebo (Placebo Comparator): Two weeks prior to the start of radiation therapy, the placebo is administered three times daily until the end of radiation therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacillus Licheniformis — Two weeks prior to the start of radiation therapy, the probiotics is administered three times daily until the end of radiation therapy.
  Other Names: Biscanen cap.
  Arms: Probiotics
Drug: Placebo — Two weeks prior to the start of radiation therapy, the placebo is administered three times daily until the end of radiation therapy.
  Other Names: Placebo oral tablet
  Arms: Placebo

SUMMARY:
In recent studies, a radiation-induced enteropathy is being reported over 50%. In clinics, probiotics are actively prescribed as a treatment for radiation-induced enteropathy. If probiotics can be used during radiation therapy to prevent or reduce radiation-induced enteropathy, the investigators can 1) reduce the inconvenience which is caused from intestinal toxicity, 2) reduce the unnecessary interruption of radiation therapy, and 3) expect to improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven uterine cancer, ovarian cancer, vaginal cancer, vulvar cancer, ureter cancer, kidney cancer, urethral cancer, and prostate cancer
* Over 20 years of age
* Eastern Cooperative Oncology Group (ECOG) score 0-2
* Appropriate values of blood test within 6 months after enrollment Absolute neutrophil count (ANC) ≥ 1500 cells/mm3, platelets≥50000cells/mm3
* Appropriate values of kidney function within 6 months after enrollment Creatinin < 2.0 ng/dL
* Appropriate values of liver function within 6 months after enrollment Total bilirubin < 1.5 times upper limit normal range, alanine aminotransferase or aspartate aminotransferase < 2.5 times upper limit normal range.
* Willing to provide informed written consent

Exclusion Criteria:

* History of pelvic irradiation
* Double primary cancer other than skin/thyroid cancer
* Combined serious morbidity
* Experience of other clinical trial within 1 month.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with grade 2 or more acute intestinal toxicities | Adverse effect evaluated at 3 months after radiation therapy
  Evaluation using CTCAE version 4.0

SECONDARY OUTCOMES:
Number of participants with grade 2 or more chronic intestinal toxicities | Adverse effect occured after 3 months since end of radiation therapy
  Evaluation using CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Young Seok Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jo YY, Kim YJ, Lee SH, Kim YS. Prevention of Radiotherapy-Induced Enteropathy by Probiotics (PREP): Double-Blind Randomized Placebo-Controlled Trial. Curr Oncol. 2024 Oct 1;31(10):5889-5895. doi: 10.3390/curroncol31100438. PMID 39451742
- [Derived] Kim YJ, Yu J, Park SP, Lee SH, Kim YS. Prevention of radiotherapy induced enteropathy by probiotics (PREP): protocol for a double-blind randomized placebo-controlled trial. BMC Cancer. 2021 Sep 16;21(1):1032. doi: 10.1186/s12885-021-08757-w. PMID 34530750